CLINICAL TRIAL: NCT05724537
Title: Durability at 20 Years of Quadrangular Resection With Annular Plication for Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: DURQUAP 2017
Record Dates: First submitted 2023-01-30; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Quadrangular resection and annular plication — Mitral regurgitation is treated removing the redundant tissue of the posterior leaflet, which is then reconstructed by sutures and plicating the posterior annulus

SUMMARY:
Degenerative mitral regurgitation (MR) due to prolapse of the posterior leaflet is the most common dysfunction of the mitral valve (MV) in the Western world and is nowadays treated with a variety of surgical techniques. Quadrangular resection combined with annular plication and annuloplasty, as originally described by Carpentier, has been the standard approach for many years, before sliding/folding plasty and artificial chordae gained larger popularity.However, very few studies have been published on thevery long-term results (up to 20 years) of quadrangular resection and annular plication, often reporting only freedom from reoperation rather than from recurrent MR. This study aims to evaluate the very long-term (20 years) clinical and echocardiographic results of this approach, which was used for many years at the beginning of our mitral repair program.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Affected by mitral valve posterior leaflet prolapse/flail causing severe mitral regurgitation
* Treated with quadrangular resection of the posterior leaflet and annulus plication

Exclusion Criteria:

* Other patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by degenerative MR, due to prolapse/flail of the posterior leaflet, treated with quadrangular resection of the posterior leaflet and annular plication
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2019-02-23 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No